CLINICAL TRIAL: NCT06005818
Title: Molecular Residual Disease (MRD) Guided Adjuvant ThErapy in Renal Cell Carcinoma (RCC)
Acronym: MRD GATE RCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Charles Peyton, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAB2369
Record Dates: First submitted 2023-08-14; First posted 2023-08-23 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Renal Cell Carcinoma
Keywords: ADJUVANT
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: MRD negative patients (No Intervention)
- Arm 2 MRD positive patients (Active Comparator): Patients are treated with Pembrolizumab 400 mg IV q 6 weeks for a total of 1 year
  Interventions: Drug: Pembrolizumab injection

INTERVENTIONS:
Drug: Pembrolizumab injection — PD-1 antibody
  Arms: Arm 2 MRD positive patients

SUMMARY:
The goal of this Clinical Study is to understand the outcomes by informing therapy choice for adjuvant treatment in clear cell renal cell carcinoma by using molecular residual disease.

The main question[s] it aims to answer are:

* what is the progression free survival of a cohort of high risk resected RCC patients when treated based on MRD
* what is the overall survival of high risk resected RCC patients when treated based on MRD

Participants will forgo adjuvant therapy with pembrolizumab if they have no detectable molecular residual disease. Participants will continue on with standard of care pembrolizumab if they do appear to have molecular residual disease.

DETAILED DESCRIPTION:
This is a multicenter open label biomarker integral treatment de-escalation study, where patients with localized renal cell carcinoma who are otherwise eligible to receive standard of care pembrolizumab will be offered observation only, if they do not demonstrate presence of molecular residual disease.

Primary Objective(s):

Provide an estimate for the 1 year -Disease-Free Survival (DFS) Provide an estimate for overall Survival (OS) for patients treated based on MRD information.

Estimate the safety of an MRD based strategy of adjuvant therapy in RCC

Primary Endpoint(s) :

i. Disease Free Survival (DFS) by Investigator's assessment as defined by RECIST 1.1

Secondary Endpoint:

i. Overall Survival at 1 year from surgery ii. Safety as defined by incidence of adverse events per NCI CTCAE v5.0

100 patients with non-metastatic clear cell renal cell carcinoma who undergo surgery to remove tumor will be enrolled, patients will be adults (≥18 years), there are no gender, age, demographic group related constraints, the trial will be conducted at centers based in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all the following criteria apply.

Type of Participant and Disease Characteristics

1. Must have histologically confirmed diagnosis of RCC with clear cell component with or without sarcomatoid features. Diagnosis of RCC with clear cell component is to be made by the investigator and does not require central histology review.

   Molecular Residual Disease
2. Patients must have at least ONE available assessment of molecular residual disease by the Signatera® (Natera Inc.) assay performed within the last 90 days prior to enrollment in study.

   Demographics
3. Be ≥18 years of age on the day of signing informed consent.

   Female Participants:
4. Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to randomization. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
5. Female participants of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of study drug.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.

   Male Participants:
6. Male participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of trial therapy through 120 days after the last dose of study therapy.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.

   Informed Consent
7. The participant provides written informed consent for the trial. The participant may also provide consent for Future Biomedical Research; however, the participant may participate in the main trial without participating in Future Biomedical Research.

   Other Inclusion Criteria
8. Have intermediate-high risk, high risk RCC as defined by the following pathological tumor-node-metastasis and Fuhrman grading status {Oza, 2022 #4431}

   1. Intermediate-high risk RCC

      * pT2, Gr. 4 or sarcomatoid, N0, M0
      * pT3, Any Gr., N0, M0
   2. High risk RCC

      * pT4, Any Gr. N0, M0
      * pT Any stage, Any Gr., N+, M0
9. Have received no prior systemic therapy for advanced RCC unless having recently initiated immunotherapy with pembrolizumab for no more than 6 weeks or 1 dose prior to enrollment.
10. Have undergone a partial nephroprotective or radical complete nephrectomy)
11. Must have undergone a nephrectomy ≥28 days prior to signing informed consent and ≤12 weeks prior to enrollment.
12. Must be tumor free as assessed by the investigator and validated by either CT or MRI scan of the brain and CAP ≤28 days from randomization.
13. Have an ECOG PS ≤2.
14. Have adequate organ function

Exclusion Criteria:

* Medical Conditions

  1. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment.
  2. Has an active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
  3. Has a known additional malignancy that is progressing or required active treatment ≤3 years ago. Exceptions include early-stage cancers (carcinoma in situ or Stage 1) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, in situ prostate cancer, or in situ breast cancer that has undergone potentially curative therapy.
  4. Has an active infection requiring systemic therapy.
  5. Has a history of, or is currently on, dialysis.
  6. Has a known history of human immunodeficiency virus infection. No human immunodeficiency virus testing is required unless mandated by local health authority.
  7. Has a known active hepatitis B (hepatitis B surface antigen reactive) or HCV (eg, HCV RNA [qualitative] is detected).
  8. Has a known history of active tuberculosis (Bacillus tuberculosis).
  9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
  10. Has a known psychiatric or substance abuse disorder that would interfere with the cooperation with the requirements of the trial in the opinion of the investigator.
  11. Has had a prior solid organ transplant.
  12. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients (refer to Investigator's Brochure for further details on excipients).
  13. A Woman of Childbearing Potential (WOCBP) who has a positive urine pregnancy test within 72 hours before randomization. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Participants must be excluded/discontinued from the trial in the event of a positive or borderline positive test result.
  14. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the Screening visit through 120 days after the last dose of study treatment.

      Prior/Concomitant Therapy
  15. Has received prior anticancer therapy and not recovered from AEs due to previously administered agents. Note: denosumab may be allowed for bone protective purposes if dosing has been stable for ≥2 weeks before screening.
  16. Has received a live vaccine within 30 days prior to the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.

      Prior/Concurrent Clinical Study Experience
  17. Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) by Investigator's assessment as defined by RECIST 1.1 | 1 year from surgery

SECONDARY OUTCOMES:
Overall Survival (OS) | 1 year from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Peyton, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided